CLINICAL TRIAL: NCT02312232
Title: Pharmacokinetics of Levodopa, Carbidopa, 3-OMD and ODM-104 After Repeated Doses of Different Formulations: an Open, Randomised, Multicentre Study With Crossover Design in Healthy Males
Brief Title: Pharmacokinetic Study in Healthy Males
Acronym: NOCOF
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3112002
Record Dates: First submitted 2014-12-02; First posted 2014-12-09 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2015-02

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Levodopa; Carbidopa; carbidopa, levodopa drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Levodopa formulation A (Experimental): Levodopa formulation A together with ODM-104 100 mg and carbidopa
  Interventions: Drug: levodopa, carbidopa, ODM-104
- levodopa formulation B (Experimental): levodopa formulation B together with ODM-104 100 mg and carbidopa
  Interventions: Drug: levodopa, carbidopa, ODM-104
- levodopa formulation C (Experimental): levodopa formulation C together with ODM-104 100 mg and carbidopa
  Interventions: Drug: levodopa, carbidopa, ODM-104
- Sinemet IR 100/25 mg (Active Comparator): Sinemet IR 100/25 mg together with ODM-104 100 mg
  Interventions: Drug: levodopa, carbidopa, ODM-104
- Half Sinemet CR 100/25 mg (Active Comparator): Half Sinemet CR 100/25 mg together with ODM-104 100 mg
  Interventions: Drug: levodopa, carbidopa, ODM-104

INTERVENTIONS:
Drug: levodopa, carbidopa, ODM-104
  Other Names: Sinemet

SUMMARY:
The purpose of this study is to investigate the pharmacokinetics of levodopa, carbidopa, 3-OMD and ODM-104 after repeated doses of 3 levodopa formulations given in combination with carbidopa and ODM-104.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent (IC) obtained.
* Good general health ascertained by detailed medical history and physical examinations.
* Finnish speaking males 18-65 years of age (inclusive).
* Normal weight defined as a body mass index (BMI) > 19 and < 32 kg/m2 (BMI = weight/height2).
* Weight at least 60 kg.
* Regular intestinal transit (no recent history of recurrent constipation, diarrhoea, or other intestinal problems).
* Participants with female partners of child-bearing potential must adhere to a proper form of contraception (hormonal contraception or intrauterine device on female partner, and an additional barrier method used at least by one of the partners) from the first study treatment administration until 3 months after the end-of-study visit.

Exclusion Criteria:

* Evidence of clinically significant cardiovascular, renal, hepatic, haematological, gastrointestinal, pulmonary, metabolic-endocrine, malignancy, neurological or psychiatric disease within the previous 2 years.
* Inherited or family history (parents, siblings) of clinically significant cardiac conduction disease.
* Current/history of inflammatory bowel disease (IBDs): Colitis ulcerosa and Crohn's disease, celiac disease. Acute duodenal or gastric ulcer or gastritis, esophagitis, colon polyps or anal fissure.
* Any condition requiring regular concomitant treatment (including vitamins and herbal products) or likely to need any concomitant treatment during the study. As an exception, paracetamol for occasional pain is allowed.
* Intake of any medication that could affect the outcome of the study.
* Any clinically significant abnormal laboratory value or physical finding (including ECG and vital signs) that in the opinion of the investigator may interfere with the interpretation of study results or constitute a health risk for the subject if he takes part in the study.
* Known hypersensitivity to the active substances or the excipients of the drugs.
* History of vasovagal collapses or vagal reactions with unexplained reason within 2 years or a tendency for vasovagal reactions during blood sampling.
* History of sleep apnea.
* Heart rate (HR) < 40 bpm or > 90 bpm after 10 minutes in supine position at the screening visit and predose.
* At the screening visit:

systolic blood pressure (BP) < 90 mmHg or > 150 mmHg after 10 minutes in supine position diastolic BP < 50 mmHg or > 90 mmHg after 10 minutes in supine position

* Abnormal 24-hour Holter findings of clinical relevance according to cardiologist´s assessment at the screening visit.
* History of anaphylactic/anaphylactoid reactions.
* History of seizures excluding febrile seizures during the first 6 years of life.
* Strong tendency to motion sickness.
* Recent or current (suspected) drug abuse.
* Recent or current alcohol abuse; regular drinking of more than 21 units per week (1 unit = 4 cl spirits or equivalent).
* Current use of nicotine containing products more than 5 cigarettes (or equivalent)/day and/or inability to refrain from the use of nicotine containing products during the study (from the screening visit to the end-of-study visit).
* Use of caffeine containing beverages more than 600 mg of caffeine/day and/or inability to refrain from the use of caffeine containing beverages during the treatment periods until 24 hours after study treatment administration.
* Blood donation or loss of significant amount of blood within 90 days prior to the first study treatment administration.
* Administration of another investigational drug within 90 days prior to the first study treatment administration.
* Unsuitable veins for repeated venipuncture or for cannulation.
* Predictable poor compliance or inability to communicate well with the study centre personnel.
* Inability to participate in all treatment periods.
* Participation in a clinical drug study during or within 3 months prior to the first study treatment administration.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-11; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (Cmax) of levodopa | 24 hours
  Peak Plasma Concentration (Cmax)

SECONDARY OUTCOMES:
Pharmacokinetics (Cmax) of carbidopa, 3-OMD and ODM-104 | 24 hours
  Peak Plasma Concentration (Cmax)

CONTACTS AND LOCATIONS:
Overall Officials: Mika Scheinin, MD, Principal Investigator — CRST Turku
Locations (1):
- CRST, Turku, Finland